CLINICAL TRIAL: NCT04374903
Title: Hydroxychloroquine in Combination With Sirolimus and Dexamethasone for Treating COVID-19 PatiEnts: A Pilot, Multicenter Randomized Open-Label Trial
Brief Title: Hydroxychloroquine in Combination With Sirolimus and Dexamethasone for Treating COVID-19 Patients
Acronym: COVID19-HOPE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study could not be implemented at the site
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Iyad Sultan, Chairman- Department of Pediatrics, Pediatrics Administration, King Hussein Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20 KHCC 74
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Patients
Keywords: COVID-19; Hydroxychloroquine; Sirolimus; Azithromycin; HOPE
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Subjects who are enrolled in the study will be randomly assigned to any of the study arms, A or B
  Study Arm A (HCQ & AZ): Subjects will receive HCQ 600mg PO X 10 days and AZ PO 250mg DAILY X 10 days.
  Study Arm B (HCQ+SIR): Subjects will receive HCQ 600mg PO X 10 days and SIR 4mg PO X 1 day then 2mg PO DAILY X 9 days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm A (HCQ & AZ) (Experimental): Subjects will receive HCQ 600mg PO X 10 days and AZ PO 250mg DAILY X 10 days.
  Interventions: Drug: HCQ & AZ vs HCQ+SIR
- Study Arm B (HCQ+SIR) (Experimental): Subjects will receive HCQ 600mg PO X 10 days and SIR 4mg PO X 1 day then 2mg PO DAILY X 9 days
  Interventions: Drug: HCQ & AZ vs HCQ+SIR

INTERVENTIONS:
Drug: HCQ & AZ vs HCQ+SIR — Subjects will receive either Hydroxychloroquine with Azithromycin or Hydroxychloroquine with Sirolimus
  Other Names: Hydroxychloroquine+Azithromycin; Hydroxychloroquine+Sirolimus

SUMMARY:
COVID-19 caused an unprecedented international crisis. There is an urgent need for an effective regimen to cure this illness. Anecdotal data and some prospective results suggested a role of antimalarial drugs (chloroquine and hydroxychloroquine) in the treatment of this disease with best available data showing value of adding azithromycin. Based on drug repurposing studies done by our team and others, we identified the autophagy/apoptosis pathway as a major target for intervention. Based on in-silico and in-vitro models, sirolimus was identified as the drug that deserves urgent prioritization. The rational for combining sirolimus and hydroxychloroquine is explained in details in the study background below and a short video prepared by study PI (https://youtu.be/-zlOMXJp2hg). The evidence for using sirolimus for influenza is emphasized by a RCT that showed reduction of mechanical ventilation time by 50% (7 days on sirolimus arm vs 15 days on oseltamivir/steroids arm). Safe administration in human subjects is illustrated by multiple phase I/II clinical trials, performed in patients with cancer. COVID19-HOPE trial will randomize patients to 2 arms: HCQ/AZ (Arm A) and HCQ/SIR (Arm B). The main inclusion criteria is an RT-PCR test confirming infection with SARS-CoV-2 along with objective clinical criteria of disease (fever, tachypnea and/or hypoxemia). The primary endpoint of study will be Time To Clinical Improvement (TTCI), defined as time from randomization to resolution of the clinical features mentioned above (no fever, no tachypnea and no hypoxemia). In addition, secondary endpoints will include clinical failure by day 28 (need for intubation and/or death), QT interval prolongation, and adverse events. The estimated NNT based on Wilcoxon Mann Whitney comparison of TTCI in study arms is 58 patients (29 each arm). The study includes an adaptive plan, meaning that after different time points the study results will be evaluated and the NNT and randomization scheme (1:1 vs. others) will be evaluated and submitted to the IRB. Also, if one arm proves to be of no value, another regimen might be introduced based on available data. The study will recruit patients for a year and once approved by IRB and JFDA attempts to recruit other centers will be made (including national and regional centers).

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female patients 18 years of age or older
* Positive RT-PCR for SARS-CoV-2.
* Fever (oral T≥39 C within 24 hours of enrollment), Tachypnea (resting respiratory rate ≥ 28/min) and/or Oxygen saturation (Sao2) ≤ 93% on room air.
* Ability to read, understand and sign IRB approved informed consent
* Patients on HCQ or HCQ/AZ already are eligible for randomization.

Exclusion Criteria:

* Weight < 40 kg.
* Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at the screening.
* Subjects with a history of retinopathy, sickle cell disease or trait, psoriasis, porphyria, history of splenectomy, mental illness or uncontrolled seizures disorder, liver cirrhosis, end-stage renal disease or need for renal replacement therapy, Decompensated heart failure, known active tuberculosis or history of incompletely treated tuberculosis, uncontrolled systemic bacterial or fungal infections, active viral infection other than COVID-19, Patients on chronic immunosuppression for other medical conditions such as rheumatological disorders, inflammatory bowel disease, or in patients with organ transplants.
* Allergy to any of the study medications.
* Drug-Drug interaction (after consulting with study PI). For example:

  * Drugs that may interact and alter HCQ level: ampicillin, cimetidine, digoxin, statins, cyclosporine, warfarin, fluconazole, within 2 weeks of dosing start, and during the duration of the study.
  * Drugs that may interact and alter SIR level: rifampicin, azole antifungals, phenytoin, diltiazem, verapamil, nicardipine, phenobarbital, carbamazepine, within 2 weeks of dosing start, and during the duration of the study.
* Any abnormal baseline laboratory screening tests listed below (Exceptions by study PI may apply if reason explained)
* Liver Child-Pugh grade C (table is included in the study)
* Creatinine >1.5 mg/dl.
* Hemoglobin for males <12 g/dl and females <10 g/dl.
* Platelet count of <100 X 103/L.
* Cardiac assessment:
* Patients with baseline corrected QT >450 msec.
* Patients with decompensated heart failure or acute myocardial infarction within the past 30 days of infection.
* Patients with HypoKalemia (<3.5 mg/dl), HypoCalcemia (<8.0 mg/dl), HypoMagnesemia (<1.6mg/dl) will be included after correction.
* Advanced respiratory support (high flow oxygen ≥ 15 L/min, CPAP, non-invasive or invasive mechanical ventilation)
* Any other significant finding based on the judgment of the PI would increase the risk of having an adverse outcome from participating in this study.
* Patients that lack decision-making capacity will not be approached to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Time to Clinical improvement (TTCI) | 28 Days
  Time to clinical improvement (TTCI), defined as time from randomization to clinical improvement, defined as resolution of fever (oral T<38), respiratory rate(<24/min) and normalization of oxygen saturation (persistent pO2 ≥95% on RA). Assessment of clinical improvement should be confirmed on 2 consecutive days in patients who do not develop clinical failure. This outcome will be analyzed separately from clinical failure (i.e. patients with clinical failure will be excluded from TTCI calculation).

SECONDARY OUTCOMES:
Clinical failure defined as death or need for Intubation and mechanical ventilation | 28 Days
  Proportion of patients who develop clinical failure, defined as death or need for mechanical ventilation within 28 days of enrollment or until discharge (whichever later).
Adverse effects | 28 Days
  Safety and tolerability, as assessed by the occurrence of adverse events in any of the study arms.
QT interval prolongation | 28 Days
  Any clinically significant increase of QT, defined as increased to over 500, or increase by 60 msec (putting the patient in over 450 msec). Proportion of patients with clinically significant increase will be used as an Outcome.
Failure to continue assigned therapy | 28 Days
  Proportion of patients who do not continue on assigned therapy will be calculated. Causes of failure to continue (drop-out) will be captured as well.
Time to viral clearance | 28 Days
  Viral RT-PCR will be performed per institutional guidelines. The time from randomization to first negative test (Which is not followed by a positive test) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided